CLINICAL TRIAL: NCT05710120
Title: Hepatitis C Screening: HCV Risk Score Alerts in CHORUS™
Brief Title: Hepatitis C Screening Alerts
Status: Completed | Type: Observational
Sponsor: Epividian (Industry)
Collaborators: Gilead Sciences (Industry); ZS (Industry); AIDS Healthcare Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: COL2023-002
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before Period (January 2022 to October 2022): All AIDS Healthcare Foundation Healthcare Centers will be contributing to the before phase of this study. In the before phase, alerts identifying patients who are eligible to be screened for hepatitis C infection will NOT be disseminated to healthcare providers and clinic staff. Routine clinical care will be administered without knowledge of the intervention.
  Interventions: Other: Standard of Care
- After Period (January 2023 to October 2023): All AIDS Healthcare Foundation Healthcare Centers will be contributing to the after phase of this study. In the after phase, alerts identifying patients who are are eligible to be screened for hepatitis C infection will be disseminated to healthcare providers and clinic staff.
  Interventions: Other: Hepatitis C Screening Alerts in CHORUS™

INTERVENTIONS:
Other: Hepatitis C Screening Alerts in CHORUS™ — ZS Associates developed a machine learning-based model that provides a numeric % chance of returning a positive hepatitis C test for a patient without diagnosed hepatitis C infection. The data used to develop the model included a US-based large scale data source including electronic medical records, medical claims, and pharmacy claims as well as social determinants of health identified from open-source data.
  Clinical Health Outcomes Reporting & Utilization Service (CHORUS™) is a web-based reporting solution that transforms electronic health record data into meaningful information for healthcare providers. CHORUS™ generates a weekly email report that alerts clinics to patients who have a scheduled appt in the coming week and may require attention. In the after period of this study, the alert will identify patients who are eligible to be screened for hepatitis C infection and provide the % chance of returning a positive hepatitis C infection test.
  Groups: After Period (January 2023 to October 2023)
Other: Standard of Care — CHORUS™ is a service provided to participating clinics and has been used by AIDS Healthcare Foundation for normal healthcare operations for quality improvement and retention in care in recent years. NO alerts identifying patients who are eligible to be screening for hepatitis C infection will be disseminated.
  Groups: Before Period (January 2022 to October 2022)

SUMMARY:
The objective of this study is to evaluate whether alerts that identify patients without hepatitis C infection to healthcare providers and clinic staff can increase the uptake of screening for hepatitis C. A period of time without alerts will be compared to a period of time with alerts.

DETAILED DESCRIPTION:
An estimated 2.4 million people in the United States were living with hepatitis C virus (HCV) infection during the period of 2013-2016. There were 4,798 new cases of acute HCV infection reported to the Centers for Disease Control (CDC) in 2020, but under ascertainment and underreporting of cases suggests that this number is less than 10% of all new HCV infections; as such, there were an estimated 66,700 new cases in 2020.

One-time screening is recommended by both the CDC and the United States Preventive Services Task Force for asymptomatic adults (aged ≥18 years and 18-79 years, respectively). The American Association for the Study of Liver Diseases and the Infectious Diseases Society of America additionally recommends annual testing for people who inject drugs and for HIV-infected men who have sex with men. Unfortunately, HCV screening rates remain low. The objective of this before and after study is to evaluate if an HCV screening algorithm, disseminated as risk score alerts in the CHORUS™ Disease Management and Clinical Considerations Report to healthcare providers and clinic staff, increases the uptake of HCV screening among patients who are HCV screening-eligible (i.e., not known to have current or prior HCV infection).

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* In care at an AIDS Healthcare Foundation Healthcare Center
* HCV screening eligible

Individuals who are HCV screening eligible include:

* HCV unknown: Never received an HCV antibody, RNA, or genotype test
* Previously HCV negative, high-risk for HCV infection: HIV-infected men who have sex with men or people who inject drugs with ≥ 1 prior negative HCV antibody or RNA test(s) who have not been screened in the prior 12 months

Exclusion Criteria:

* <18 years of age
* Diagnosed HCV infection (i.e., reactive HCV antibody, detectable HCV RNA test, or HCV genotype test)

Individuals with diagnosed HCV infection include:

* Acute HCV infection, untreated or in treatment
* Chronic HCV infection, untreated or in treatment
* Spontaneous clearance of prior HCV infection
* Sustained virologic response after direct acting antiviral therapy for prior HCV infection
* Treatment failure after direct acting antiviral therapy for prior HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic Population: AIDS Healthcare Foundation Healthcare Centers across the United States and Puerto Rico are included in the study.
  Patient Population: Adult patients without diagnosed HCV infection who are HCV screening eligible at AIDS Healthcare Foundation Healthcare Centers are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 125706 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Screening to Diagnosis Ratio for Hepatitis C Infection | End of follow-up (Before study period: October 2022; After study period: October 2023)
  Number of HCV screening-eligible individuals who complete a visit and who are screened by either an HCV antibody or HCV RNA test divided by the number of individuals whose HCV RNA test returns a detectable result (i.e., people with active HCV infection).

SECONDARY OUTCOMES:
Screening Tests for Hepatitis C Infection | End of follow-up (Before study period: October 2022; After study period: October 2023)
  Proportion of HCV screening-eligible patients who receive HCV antibody test alone, HCV RNA test alone, and reactive HCV antibody test followed by an HCV RNA or genotype test.
HCV RNA Viral Load Tests | End of follow-up (Before study period: October 2022; After study period: October 2023)
  Among individuals who screen positive for HCV infection (i.e., reactive HCV antibody test) over follow-up, the distribution of HCV RNA test results (i.e., detectable, not detectable)
HCV Screening History | Baseline (Before study period: January 2022; After study period: January 2023)
  The HCV screening history for HCV screening-eligible individuals who were previously HCV negative but are at high-risk for HCV infection (i.e., HIV-infected men who have sex with men and people who inject drugs) will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Dieterich, MD, Principal Investigator — Mount Sinai Healthcare System
Locations (1):
- AIDS Healthcare Foundation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No